CLINICAL TRIAL: NCT01092247
Title: The Effect of Ketogenic Diet on Malignant Tumors- Recurrence and Progress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Nutricia Liverpool (Industry)
Responsible Party: Faith Takurukura BAppSc. PGDip.Diet. RGN, Clinical Trials Specialist, Research & Development, Nutricia Liverpool
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TASMC-09-NV-0056-CTIL
Record Dates: First submitted 2010-03-15; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-02

CONDITIONS: Malignant Tumors
Keywords: Patients with malignant tumors
MeSH Terms: conditions — Neoplasms | interventions — Nutritional Support

ARMS (2):
- Standard diet: Nutritional support (Placebo Comparator)
  Interventions: Other: Nutritional support with Standard diet
- Nutritional intervention: Ketogenic diet. (Experimental)
  Interventions: Other: Nutritional intervention with the Ketogenic diet

INTERVENTIONS:
Other: Nutritional support with Standard diet — Nutritional support with Standard diet
  Arms: Standard diet: Nutritional support
Other: Nutritional intervention with the Ketogenic diet — Nutritional intervention with ketogenic diet. The Diet plan will be based on each patient individually according to his nutritional needs. Age, weight, activity levels, culture and food preferences are taken in consideration
  Arms: Nutritional intervention: Ketogenic diet.

SUMMARY:
The aim of the study is, to study the efficacy of the ketogenic diet in delaying or preventing recurrence and tumor growth progression of patients who have been previously treated by concomitant chemoradiotherapy (6 months) for high-grade glial tumors.

It will be an open-label trial of nutritional intervention for up to 1 year. An interim analysis of the data will be carried out to assess safety, compliance and efficacy of the diet. This will be reviewed by both SHS and the Clinical trial team.

ELIGIBILITY:
Inclusion criteria:

1. Consenting adults aged ≥ 18 years.
2. Recurrent or progressive high grade glioma after failure of at least one line of standard oncological treatment.
3. Gliomatosis cerebri, including patients declining radiation treatment.

Exclusion criteria:

1. Patients with malignant tumors who are receiving treatment at the time of the recruitment.
2. Early termination - patients who will wish to stop their participation in the trial will discontinue the ketogenic diet and return to their usual diet.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-05 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
To study the effect of the ketogenic diet on tumor growth progression and longevity in patients with Malignant glioblastoma.
  This will be done by comparing tumor size by repeated MRI studies (every 2 months)

SECONDARY OUTCOMES:
Quality of life
  Performance scale and quality of life evaluation (Karnofsky and EQ5D scale)